CLINICAL TRIAL: NCT03985033
Title: The Clinical and Biological Effects of Leucocyte and Platelet-rich Fibrin (L-PRF) on Post-extraction Sockets Healing: a Randomized Controlled Trial
Brief Title: The Clinical and Biological Effects of Leucocyte and Platelet-rich Fibrin (L-PRF) on Post-extraction Sockets Healing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The European Research Group on Periodontology (ERGOPerio) (Network)
Collaborators: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Maurizio Tonetti, Executive Director, Clinical Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: HKUPhD20190528
Record Dates: First submitted 2019-06-10; First posted 2019-06-13 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2022-01

CONDITIONS: Tooth Extraction
MeSH Terms: interventions — Leukocyte Count

STUDY DESIGN:
Intervention Model Description: Split-mouth design allowing to assess two types of treatment in the same patient.
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- L-PRF (Experimental): Post-extraction sockets will be filled with autologous leucocyte and platelet-rich fibrin (L-PRF) clot.
  Interventions: Other: leucocyte and platelet-rich fibrin (L-PRF)
- Control (No Intervention): Post-extraction sockets will be left to heal spontaneously with natural blood clot.

INTERVENTIONS:
Other: leucocyte and platelet-rich fibrin (L-PRF) — The blood collected from each patient will be centrifuged immediately at 2700 rpm for 12 min to separate L-PRF.
  Arms: L-PRF

SUMMARY:
This study evaluates the clinical and biological effects of leucocyte and platelet-rich fibrin (L-PRF) on post-extraction sockets healing.

DETAILED DESCRIPTION:
Tooth extraction is one of the most frequent dental surgical procedures. Following tooth extraction, dimensional changes of the alveolus are inevitable, which consequently decrease the height and width of alveolar bone and impair ideal implant placement and conventional prosthetic treatment. In order to reduce the bone resorption after tooth extraction, the use of platelet concentrates has been proposed. Platelet rich fibrin (PRF) is a second generation of platelet concentrates consisting of platelets, leukocyte and growth factors harvested from blood. PRF not only supports hemostasis but also favors the natural wound healing process. Over the past decade, PRF has gained tremendous momentum having been utilized for a variety of dental and medical procedures including the management of post-extraction sockets. To date, several studies have assessed the efficacy of the use of PRF in promoting postextraction sockets healing. However, results remain contradictory and mainly focus on the clinical and radiological hard and soft tissue healing, aesthetics and postoperative discomfort. The mechanistic hypothesis is that growth factors released by PRF preparations modulate the wound healing process but the effect of local PRF application on the kinetics of release of wound healing modulators has not been studied so far. There is also a lack of information in the literature regarding the biological evaluation during postextraction sockets healing to understand the potential mechanisms. In order to assess the presence or follow dynamics of biomarkers, in this study wound fluid (WF) will be collected from the post-extraction sockets and utilized for multiplex immunoassay. Multiplex immunoassay allows simultaneous quantification of multiple markers providing unique information for a more complete understanding of the potential mechanism of PRF and spontaneous extraction socket healing. Therefore, the aim of this randomized clinical trial is to evaluate the effects of PRF on biomarkers response during post-extraction sockets healing.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study
* Healthy males and females of age 18-70
* Need for two or more extractions of single rooted teeth in the presence of adjacent teeth or implants due to unrestorable caries, residual roots, root fractures or orthodontic treatment
* Able (in the investigators opinion) and willing to comply with all study requirements
* Interested in tooth replacement with dental implants

Exclusion Criteria:

* Endodontic periapical lesions with a diameter of more than 5 mm (radiographically determined)
* Sites with buccal and lingual bone plate loss more than 5 mm
* Frank purulence or acute abscess at the time of extraction
* Pregnancy or lactation
* Smokers or alcoholics
* Platelet dysfunction syndrome or thrombocytopenia
* Uncontrolled diabetes
* Medical contraindications to elective oral surgery procedures

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Concentrations changes of the molecules and inflammatory mediators | Baseline, 6 hours, 24 hours, 3 days and 7 days
  Concentrations changes of the molecules and inflammatory mediators in the gingival crevicular fluid (GCF) or wound fluid (WF) from the extraction sockets in L-PRF group and control group at baseline (from GCF), 6 hours, 24 hours, 3 days, 7 days.

SECONDARY OUTCOMES:
Genes expression profiles | Baseline and 3 days
  Genes expression profiles of the growth and differentiation factors and inflammatory mediators from the tissue specimen taken from the post-extraction sockets at 3 days.
Laser Doppler Flowmetry (LDF) measurement | Before and immediately after the tooth extraction, 6 hours, 24 hours, 3 days and 7 days
  A commercially available Laser Doppler Blood FlowMeter equipped with a standard fiber optic probe will be used for LDF measurements before tooth extraction, immediately postoperatively, 6 hours, 24 hours, 3 days and 7 days.
Radiographic bone changes (Cone-beam computed tomography) | Baseline and 4 months
  Cone-beam computed tomography (CBCT) images will be obtained before extraction as the baseline and at the 4 months.
Wound Healing Index (HI) | 6 hours, 24 hours, 3 days and 7 days
  Soft tissue healing will be assessed by Wound Healing Index (1 = very poor, 2 = poor, 3 = good, 4 = very good, 5 = excellent).
Visual analog scale (VAS) | 6 hours, 24 hours, 3 days and 7 days
  A 10-point VAS with a score of 0 that equals "no pain" and a score of 10 that equals "worst pain imaginable" will be used to evaluate the postoperative pain at 6 hours, 24 hours, 3 days and 7 days. The patients will be asked to fill the pain they feel at the time of questioning. Questionnaires will be collected at the one-week follow-up visit.

CONTACTS AND LOCATIONS:
Overall Officials: Maurizio Tonetti, DMD, Principal Investigator — The European Research Group on Periodontology (ERGOPerio)
Locations (1):
- Faculty of Dentistry, The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alssum L, Eubank TD, Roy S, Erdal BS, Yildiz VO, Tatakis DN, Leblebicioglu B. Gingival Perfusion and Tissue Biomarkers During Early Healing of Postextraction Regenerative Procedures: A Prospective Case Series. J Periodontol. 2017 Nov;88(11):1163-1172. doi: 10.1902/jop.2017.170117. Epub 2017 Jun 23. PMID 28644107
- [Background] Araujo MG, Silva CO, Misawa M, Sukekava F. Alveolar socket healing: what can we learn? Periodontol 2000. 2015 Jun;68(1):122-34. doi: 10.1111/prd.12082. PMID 25867983
- [Background] Avila-Ortiz G, Chambrone L, Vignoletti F. Effect of alveolar ridge preservation interventions following tooth extraction: A systematic review and meta-analysis. J Clin Periodontol. 2019 Jun;46 Suppl 21:195-223. doi: 10.1111/jcpe.13057. Erratum In: J Clin Periodontol. 2020 Jan;47(1):129. doi: 10.1111/jcpe.13212. PMID 30623987
- [Background] Avila-Ortiz G, Elangovan S, Kramer KW, Blanchette D, Dawson DV. Effect of alveolar ridge preservation after tooth extraction: a systematic review and meta-analysis. J Dent Res. 2014 Oct;93(10):950-8. doi: 10.1177/0022034514541127. Epub 2014 Jun 25. PMID 24966231
- [Background] Buser D, Hoffmann B, Bernard JP, Lussi A, Mettler D, Schenk RK. Evaluation of filling materials in membrane--protected bone defects. A comparative histomorphometric study in the mandible of miniature pigs. Clin Oral Implants Res. 1998 Jun;9(3):137-50. doi: 10.1034/j.1600-0501.1998.090301.x. PMID 10530128
- [Background] Chan D, Pelekos G, Ho D, Cortellini P, Tonetti MS. The depth of the implant mucosal tunnel modifies the development and resolution of experimental peri-implant mucositis: A case-control study. J Clin Periodontol. 2019 Feb;46(2):248-255. doi: 10.1111/jcpe.13066. Epub 2019 Feb 7. PMID 30638273
- [Background] Del Fabbro M, Bucchi C, Lolato A, Corbella S, Testori T, Taschieri S. Healing of Postextraction Sockets Preserved With Autologous Platelet Concentrates. A Systematic Review and Meta-Analysis. J Oral Maxillofac Surg. 2017 Aug;75(8):1601-1615. doi: 10.1016/j.joms.2017.02.009. Epub 2017 Feb 20. PMID 28288724
- [Background] Franceschi RT. Biological approaches to bone regeneration by gene therapy. J Dent Res. 2005 Dec;84(12):1093-103. doi: 10.1177/154405910508401204. PMID 16304438
- [Background] Gamal AY, Abdel Ghaffar KA, Alghezwy OA. Crevicular Fluid Growth Factors Release Profile Following the Use of Platelet-Rich Fibrin and Plasma Rich Growth Factors in Treating Periodontal Intrabony Defects: A Randomized Clinical Trial. J Periodontol. 2016 Jun;87(6):654-62. doi: 10.1902/jop.2016.150314. Epub 2016 Feb 15. PMID 26876351
- [Background] Hammerle CH, Araujo MG, Simion M; Osteology Consensus Group 2011. Evidence-based knowledge on the biology and treatment of extraction sockets. Clin Oral Implants Res. 2012 Feb;23 Suppl 5:80-2. doi: 10.1111/j.1600-0501.2011.02370.x. PMID 22211307
- [Background] Jung RE, Philipp A, Annen BM, Signorelli L, Thoma DS, Hammerle CH, Attin T, Schmidlin P. Radiographic evaluation of different techniques for ridge preservation after tooth extraction: a randomized controlled clinical trial. J Clin Periodontol. 2013 Jan;40(1):90-8. doi: 10.1111/jcpe.12027. Epub 2012 Nov 19. PMID 23163915
- [Background] Kampfer H, Pfeilschifter J, Frank S. Expressional regulation of angiopoietin-1 and -2 and the tie-1 and -2 receptor tyrosine kinases during cutaneous wound healing: a comparative study of normal and impaired repair. Lab Invest. 2001 Mar;81(3):361-73. doi: 10.1038/labinvest.3780244. PMID 11310829
- [Background] Lin Z, Rios HF, Volk SL, Sugai JV, Jin Q, Giannobile WV. Gene expression dynamics during bone healing and osseointegration. J Periodontol. 2011 Jul;82(7):1007-17. doi: 10.1902/jop.2010.100577. Epub 2010 Dec 13. PMID 21142982
- [Background] Marenzi G, Riccitiello F, Tia M, di Lauro A, Sammartino G. Influence of Leukocyte- and Platelet-Rich Fibrin (L-PRF) in the Healing of Simple Postextraction Sockets: A Split-Mouth Study. Biomed Res Int. 2015;2015:369273. doi: 10.1155/2015/369273. Epub 2015 Jul 26. PMID 26273612
- [Background] Miron RJ, Zucchelli G, Pikos MA, Salama M, Lee S, Guillemette V, Fujioka-Kobayashi M, Bishara M, Zhang Y, Wang HL, Chandad F, Nacopoulos C, Simonpieri A, Aalam AA, Felice P, Sammartino G, Ghanaati S, Hernandez MA, Choukroun J. Use of platelet-rich fibrin in regenerative dentistry: a systematic review. Clin Oral Investig. 2017 Jul;21(6):1913-1927. doi: 10.1007/s00784-017-2133-z. Epub 2017 May 27. PMID 28551729
- [Background] Moraschini V, Barboza ES. Effect of autologous platelet concentrates for alveolar socket preservation: a systematic review. Int J Oral Maxillofac Surg. 2015 May;44(5):632-41. doi: 10.1016/j.ijom.2014.12.010. Epub 2015 Jan 24. PMID 25631334
- [Background] Singh A, Kohli M, Gupta N. Platelet rich fibrin: a novel approach for osseous regeneration. J Maxillofac Oral Surg. 2012 Dec;11(4):430-4. doi: 10.1007/s12663-012-0351-0. Epub 2012 Apr 10. PMID 24293936
- [Background] Srinivas B, Das P, Rana MM, Qureshi AQ, Vaidya KC, Ahmed Raziuddin SJ. Wound Healing and Bone Regeneration in Postextraction Sockets with and without Platelet-rich Fibrin. Ann Maxillofac Surg. 2018 Jan-Jun;8(1):28-34. doi: 10.4103/ams.ams_153_17. PMID 29963421
- [Background] Tan WL, Wong TL, Wong MC, Lang NP. A systematic review of post-extractional alveolar hard and soft tissue dimensional changes in humans. Clin Oral Implants Res. 2012 Feb;23 Suppl 5:1-21. doi: 10.1111/j.1600-0501.2011.02375.x. PMID 22211303
- [Background] Temmerman A, Vandessel J, Castro A, Jacobs R, Teughels W, Pinto N, Quirynen M. The use of leucocyte and platelet-rich fibrin in socket management and ridge preservation: a split-mouth, randomized, controlled clinical trial. J Clin Periodontol. 2016 Nov;43(11):990-999. doi: 10.1111/jcpe.12612. Epub 2016 Sep 21. PMID 27509214
- [Background] Tonetti M, Cugini MA, Goodson JM. Zero-order delivery with periodontal placement of tetracycline-loaded ethylene vinyl acetate fibers. J Periodontal Res. 1990 Jul;25(4):243-9. doi: 10.1111/j.1600-0765.1990.tb00911.x. PMID 2142733
- [Background] Van der Weijden F, Dell'Acqua F, Slot DE. Alveolar bone dimensional changes of post-extraction sockets in humans: a systematic review. J Clin Periodontol. 2009 Dec;36(12):1048-58. doi: 10.1111/j.1600-051X.2009.01482.x. PMID 19929956
- [Background] Werner S, Grose R. Regulation of wound healing by growth factors and cytokines. Physiol Rev. 2003 Jul;83(3):835-70. doi: 10.1152/physrev.2003.83.3.835. PMID 12843410
- [Derived] Wang X, Fok MR, Pelekos G, Jin L, Tonetti MS. Increased local concentrations of growth factors from leucocyte- and platelet-rich fibrin do not translate into improved alveolar ridge preservation: An intra-individual mechanistic randomized controlled trial. J Clin Periodontol. 2022 Sep;49(9):889-898. doi: 10.1111/jcpe.13688. Epub 2022 Jul 17. PMID 35734895